CLINICAL TRIAL: NCT01254565
Title: A Double-Blind, Randomized, Placebo-Controlled Multiple Ascending Dose Study to Assess the Safety, Tolerability and Efficacy of KAI-4169 in Hemodialysis Subjects With Secondary Hyperparathyroidism
Brief Title: Safety, Tolerability and Efficacy of Etelcalcetide in Hemodialysis Patients With Secondary Hyperparathyroidism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KAI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: KAI-4169-003; 20120330 (Other: Amgen, Inc)
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Clinical Trial, Phase 2; Renal Dialysis; Secondary Hyperparathyroidism; Parathyroid hormone
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Etelcalcetide (Experimental): Participants received etelcalcetide administered by intravenous injection at the end of each hemodialysis session three times a week (TIW). The starting dose level was 5 mg; dose escalation was to proceed to 10 and 20 mg pending safety review of the prior cohort.
  Interventions: Drug: Etelcalcetide
- Placebo (Placebo Comparator): Participants received placebo administered by intravenous injection at the end of each hemodialysis session three times a week (TIW).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etelcalcetide — Administered intravenously (IV) at the end of hemodialysis
  Other Names: KAI-4169; AMG 416; Parsabiv™
  Arms: Etelcalcetide
Drug: Placebo — Administered intravenously at the end of hemodialysis
  Arms: Placebo

SUMMARY:
The purpose of this study is to characterize the safety and tolerability and efficacy of multiple ascending doses of etelcalcetide in hemodialysis patients for the treatment of secondary hyperparathyroidism (HPT).

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent.
* Intact parathyroid hormone (PTH) at least 350 pg/mL.
* Corrected calcium at least 9.0 mg/dL.
* Hemoglobin at least 9.0 g/dL.
* Adequate hemodialysis three times per week.
* Excepting chronic renal failure, subject is judged to be in stable medical condition based on medical history, physical examination, and routine laboratory tests.

Exclusion Criteria:

* History or symptomatic ventricular dysrhythmias.
* History of angina pectoris or congestive heart failure
* History of myocardial infarction, coronary angioplasty, or coronary artery bypass grafting within the past 6 months.
* History of or treatment for seizure disorder.
* Recent (3 months) parathyroidectomy.
* Serum transaminases (alanine aminotransferase, aspartate aminotransferase) greater than two times the upper limit of normal at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-02-20; Primary Completion 2011-07 (Actual); Study Completion 2011-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M D, Study Director — Amgen
Locations (12):
- United States (12):
  - Azusa, California
  - Costa Mesa, California
  - Lynwood, California
  - Riverside, California
  - San Diego, California
  - Denver, Colorado
  - Macon, Georgia
  - Shreveport, Louisiana
  - Brooklyn Center, Minnesota
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Chesapeake, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 11 study centers in the United States from 17 February 2011 (first participant enrolled) to 24 August 2011 (last participant completed follow up). A total of 87 patients with secondary hyperparathyroidism (HPT) receiving hemodialysis were enrolled and randomized in the study.
Pre-assignment Details: This was a multiple-ascending dose study consisting of 3 cohorts: Cohort 1 participants were randomized in a 3:2 ratio to receive etelcalcetide or placebo for 2 weeks; Cohorts 2 and 3 were randomized in a 1:1 ratio to receive etelcalcetide or placebo for 4 weeks. Randomization was stratified by serum parathyroid hormone (< 600 or ≥ 600 pg/mL).
Groups:
- Cohort 1: Placebo: Participants received placebo administered by intravenous injection at the end of each hemodialysis session three times a week (TIW) for 2 weeks.
- Cohort 1: Etelcalcetide 5 mg: Participants received 5 mg etelcalcetide administered by intravenous injection at the end of each hemodialysis session TIW for 2 weeks.
- Cohort 2: Placebo; Cohort 3: Placebo: Participants received placebo administered by intravenous injection at the end of each hemodialysis session TIW for 4 weeks.
- Cohort 2: Etelcalcetide 10 mg: Participants received 10 mg etelcalcetide administered by intravenous injection at the end of each hemodialysis session TIW for 4 weeks.
- Cohort 3: Etelcalcetide 5 mg: Participants received 5 mg etelcalcetide administered by intravenous injection at the end of each hemodialysis session TIW for 4 weeks.
Period: Overall Study
Arm/Group | Cohort 1: Placebo | Cohort 1: Etelcalcetide 5 mg | Cohort 2: Placebo | Cohort 2: Etelcalcetide 10 mg | Cohort 3: Placebo | Cohort 3: Etelcalcetide 5 mg
Started | 5 | 7 | 21 | 21 | 16 | 17
Received Treatment | 4 | 6 | 21 | 21 | 13 | 13
Completed | 4 | 6 | 21 | 20 | 12 | 13
Not Completed | 1 | 1 | 0 | 1 | 4 | 4
Not completed — Non-compliance to Study Procedures | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Did not Receive Treatment | 1 | 1 | 0 | 0 | 3 | 4
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one 1 dose of investigational product (the modified intent-to-treat [mITT] population)
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Placebo | Cohort 1: Etelcalcetide 5 mg | Cohort 2: Placebo | Cohort 2: Etelcalcetide 10 mg | Cohort 3: Placebo | Cohort 3: Etelcalcetide 5 mg | Total
Number analyzed (Participants) | 4 | 6 | 21 | 21 | 13 | 13 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (16.66) | 54.0 (10.00) | 52.4 (13.65) | 50.7 (13.60) | 56.7 (11.61) | 59.6 (10.99) | 53.7 (12.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 8 | 6 | 5 | 5 | 30
  Male | 2 | 2 | 13 | 15 | 8 | 8 | 48
Race [Count of Participants; unit: Participants]
  White | 2 | 1 | 1 | 3 | 4 | 4 | 15
  Black or African American | 2 | 5 | 20 | 18 | 9 | 9 | 63
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 2 | 2 | 3 | 8
  Not Hispanic or Latino | 4 | 5 | 21 | 19 | 11 | 10 | 70
Stratification Factor: Screening Serum Parathyroid Hormone (PTH) [Count of Participants; unit: Participants]
  < 600 pg/mL | 3 | 4 | 11 | 12 | 7 | 9 | 46
  ≥ 600 pg/mL | 1 | 2 | 10 | 9 | 6 | 4 | 32
Parathyroid Hormone [Mean (Standard Deviation); unit: pg/mL] | 636.3 (191.64) | 588.3 (250.52) | 601.5 (239.20) | 765.1 (480.82) | 619.4 (310.35) | 662.1 (442.01) | 659.4 (361.28)
Corrected Calcium [Mean (Standard Deviation); unit: mg/dL] — Population: Corrected calcium data were missing for 2 participants in Cohort 3.
  mg/dL
    number analyzed (Participants) | 4 | 6 | 21 | 21 | 12 | 12 | 76
    (all) | 9.1 (0.84) | 9.3 (0.44) | 9.8 (0.62) | 9.7 (0.59) | 9.3 (0.58) | 9.7 (0.62) | 9.6 (0.63)
Phosphorus [Mean (Standard Deviation); unit: mg/dL] — Population: Phosphorus values were not collected at Baseline for Cohort 1; data were missing for 7 participants in Cohort 2 and 2 participants in Cohort 3.
  mg/dL
    number analyzed (Participants) | 0 | 0 | 18 | 17 | 12 | 12 | 59
    (all) |  |  | 6.5 (1.83) | 5.7 (1.18) | 5.2 (1.17) | 5.0 (1.02) | 5.7 (1.49)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Mean Pre-hemodialysis Parathyroid Hormone (PTH) During the Efficacy Assessment Phase
Description: Baseline is defined as the average of pre-hemodialysis values obtained on day -2 and day 1. The efficacy assessment phase (defined as 3 days before and 3 days after the last dose of investigational product) value is the mean of all predialysis values obtained during that period.
Time Frame: Baseline and the efficacy assessment phase (EAP; defined as the period between 3 days before and 3 days after the last dose of study drug; approximately 2 weeks for Cohort 1 and 4 weeks for Cohorts 2 and 3)
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1: Placebo | Cohort 1: Etelcalcetide 5 mg | Cohort 2: Placebo | Cohort 2: Etelcalcetide 10 mg | Cohort 3: Placebo | Cohort 3: Etelcalcetide 5 mg
Number analyzed (Participants) | 4 | 6 | 21 | 21 | 13 | 13
percent change | 0.3 (17.11) | -19.4 (20.65) | 28.5 (70.39) | -49.4 (20.42) | 2.3 (29.44) | -33.0 (26.28)
Statistical Analysis 1: Comparison: Cohort 2: Placebo vs Cohort 2: Etelcalcetide 10 mg; The hypothesis for this study (Cohorts 2 and 3) was that intravenous administration of etelcalcetide is superior to placebo for the reduction of PTH after TIW dosing in hemodialysis patients with secondary HPT. This hypothesis was tested in Cohorts 2 and 3 by comparing the mean percent changes from baseline in pre-hemodialysis PTH levels collected during the efficacy phase between the etelcalcetide and placebo groups within each cohort; Test type: Superiority — The primary endpoint was tested at the 0.05 level (1-sided); p < 0.0001, ANOVA; A rank analysis of variance (ANOVA) model with treatment and screening PTH (< 600 pg/mL or ≥ 600 pg/mL) as factors; LS Mean Difference = -76.9, 95% CI 2-sided [-86.9 to -50.0]
Statistical Analysis 2: Comparison: Cohort 3: Placebo vs Cohort 3: Etelcalcetide 5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The primary endpoint was tested at the 0.05 level (1-sided); p = 0.0032, ANOVA; ANOVA model with treatment and screening PTH (< 600 pg/mL or ≥ 600 pg/mL) as factors; LS Mean Difference = -36.7, 95% CI 2-sided [-59.8 to -13.6]

2. Secondary Outcome: Percentage of Participants With ≥ 30% Reduction From Baseline in Mean Parathyroid Hormone During the Efficacy Assessment Phase
Description: as for outcome 1
Time Frame: Baseline and the efficacy assessment phase (from 3 days before to 3 days after the last dose of study drug; approximately 2 weeks for Cohort 1 and 4 weeks for Cohorts 2 and 3)
Population: Modified intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Etelcalcetide 5 mg | Cohort 2: Placebo | Cohort 2: Etelcalcetide 10 mg | Cohort 3: Placebo | Cohort 3: Etelcalcetide 5 mg
Number analyzed (Participants) | 4 | 6 | 21 | 21 | 13 | 13
percentage of participants | 0.0 | 33.3 | 9.5 | 76.2 | 15.4 | 53.8
Statistical Analysis 1: Comparison: Cohort 2: Placebo vs Cohort 2: Etelcalcetide 10 mg; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 2: Comparison: Cohort 3: Placebo vs Cohort 3: Etelcalcetide 5 mg; Test type: Superiority; p = 0.0968, Fisher Exact

3. Secondary Outcome: Percentage of Participants With Mean Parathyroid Hormone ≤ 300 pg/mL During the Efficacy Assessment Phase
Description: The efficacy assessment phase (defined as 3 days before and 3 days after the last dose of investigational product) value is the mean of all predialysis values obtained during that period.
Time Frame: Efficacy assessment phase (from 3 days before to 3 days after the last dose of study drug; approximately 2 weeks for Cohort 1 and 4 weeks for Cohorts 2 and 3)
Population: Modified intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Etelcalcetide 5 mg | Cohort 2: Placebo | Cohort 2: Etelcalcetide 10 mg | Cohort 3: Placebo | Cohort 3: Etelcalcetide 5 mg
Number analyzed (Participants) | 4 | 6 | 21 | 21 | 13 | 13
percentage of participants | 0.0 | 16.7 | 4.8 | 66.7 | 7.7 | 46.2
Statistical Analysis 1: Comparison: Cohort 2: Placebo vs Cohort 2: Etelcalcetide 10 mg; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 2: Comparison: Cohort 3: Placebo vs Cohort 3: Etelcalcetide 5 mg; Test type: Superiority; p = 0.0730, Fisher Exact

4. Secondary Outcome: Percent Change From Baseline in Mean Corrected Calcium (cCa) During the Efficacy Assessment Phase
Description: as for outcome 1
Time Frame: as for outcome 2
Population: Modified intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1: Placebo | Cohort 1: Etelcalcetide 5 mg | Cohort 2: Placebo | Cohort 2: Etelcalcetide 10 mg | Cohort 3: Placebo | Cohort 3: Etelcalcetide 5 mg
Number analyzed (Participants) | 4 | 6 | 21 | 21 | 12 | 12
percent change | 1.7 (3.76) | -7.3 (2.62) | -1.7 (6.25) | -13.0 (10.17) | 1.0 (5.26) | -6.0 (7.95)
Statistical Analysis 1: Comparison: Cohort 2: Placebo vs Cohort 2: Etelcalcetide 10 mg; Test type: Superiority; p < 0.0001, ANOVA; A rank ANOVA model with treatment and screening PTH (< 600 or ≥ 600 pg/mL) as factors; LS Mean Difference = -11.3, 95% CI 2-sided [-16.4 to -8.4]
Statistical Analysis 2: Comparison: Cohort 3: Placebo vs Cohort 3: Etelcalcetide 5 mg; Test type: Superiority; p = 0.0235, ANOVA; ANOVA model with treatment and screening PTH (< 600 or ≥ 600 pg/mL) as factors; LS Mean Difference = -6.9, 95% CI 2-sided [-12.8 to -1.0]

5. Secondary Outcome: Percent Change From Baseline in Mean Phosphorus (P) During the Efficacy Assessment Phase
Description: as for outcome 1
Time Frame: as for outcome 2
Population: Modified intent-to-treat population with available data; Phosphorus data were not collected at baseline for participants in Cohort 1.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1: Placebo | Cohort 1: Etelcalcetide 5 mg | Cohort 2: Placebo | Cohort 2: Etelcalcetide 10 mg | Cohort 3: Placebo | Cohort 3: Etelcalcetide 5 mg
Number analyzed (Participants) | 0 | 0 | 17 | 17 | 12 | 12
percent change |  |  | 1.4 (17.92) | -2.4 (26.86) | 14.1 (36.05) | -7.3 (12.83)
Statistical Analysis 1: Comparison: Cohort 2: Placebo vs Cohort 2: Etelcalcetide 10 mg; Test type: Superiority; p = 0.2255, ANOVA; A rank ANOVA model with treatment and screening PTH (< 600 or ≥ 600 pg/mL) as factors; LS Mean Difference = -4.2, 95% CI 2-sided [-18.6 to 5.7]
Statistical Analysis 2: Comparison: Cohort 3: Placebo vs Cohort 3: Etelcalcetide 5 mg; Test type: Superiority; p = 0.1751, ANOVA; A rank ANOVA model with treatment and screening PTH (< 600 or ≥ 600 pg/mL) as factors; LS mean Difference = -21.8, 95% CI 2-sided [-29.8 to 5.9]

6. Secondary Outcome: Percent Change From Baseline in Corrected Calcium Phosphorus Product (cCa x P) During the Efficacy Assessment Phase
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1: Placebo | Cohort 1: Etelcalcetide 5 mg | Cohort 2: Placebo | Cohort 2: Etelcalcetide 10 mg | Cohort 3: Placebo | Cohort 3: Etelcalcetide 5 mg
Number analyzed (Participants) | 0 | 0 | 17 | 17 | 12 | 12
percent change |  |  | -0.3 (16.25) | -11.0 (32.32) | 14.7 (35.79) | -12.6 (14.99)
Statistical Analysis 1: Comparison: Cohort 2: Placebo vs Cohort 2: Etelcalcetide 10 mg; Test type: Superiority; p = 0.0112, ANOVA; A rank ANOVA model with treatment and screening PTH (< 600 or ≥ 600 pg/mL) as factors; LS Mean Difference = -11.2, 95% CI 2-sided [-26.8 to -4.9]
Statistical Analysis 2: Comparison: Cohort 3: Placebo vs Cohort 3: Etelcalcetide 5 mg; Test type: Superiority; p = 0.0554, ANOVA; A rank ANOVA model with treatment and screening PTH (< 600 or ≥ 600 pg/mL) as factors; LS Mean Difference = -27.7, 95% CI 2-sided [-39.3 to -1.6]

7. Secondary Outcome: Percentage of Participants With Mean Phosphorus ≤ 4.5 mg/dL or ≤ 5.5 mg/dL During the Efficacy Assessment Phase
Time Frame: Efficacy assessment phase
Population: Modified intent to treat population
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: Etelcalcetide 5 mg | Cohort 2: Placebo | Cohort 2: Etelcalcetide 10 mg | Cohort 3: Placebo | Cohort 3: Etelcalcetide 5 mg
Number analyzed (Participants) | 4 | 6 | 21 | 21 | 13 | 13
percentage of participants
  Phosphorus ≤ 4.5 mg/dL | 0.0 | 0.0 | 4.8 | 47.6 | 15.4 | 46.2
  Phosphorus ≤ 5.5 mg/dL | 0.0 | 0.0 | 33.3 | 66.7 | 53.8 | 76.9

ADVERSE EVENTS:
Time Frame: From first dose of study drug through to day 41 (Cohort 1) or day 55 (Cohorts 2 and 3).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Cohort 1: Placebo: Participants received placebo administered by intravenous injection at the end of each hemodialysis session TIW for 2 weeks.
Arm/Group | Cohort 1: Placebo | Cohort 1: Etelcalcetide 5 mg | Cohort 2: Placebo | Cohort 2: Etelcalcetide 10 mg | Cohort 3: Placebo | Cohort 3: Etelcalcetide 5 mg
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/6 | 2/21 | 3/21 | 1/13 | 3/13
Other Adverse Events (participants affected / at risk) | 1/4 | 4/6 | 5/21 | 2/21 | 2/13 | 3/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Placebo (N=4) | Cohort 1: Etelcalcetide 5 mg (N=6) | Cohort 2: Placebo (N=21) | Cohort 2: Etelcalcetide 10 mg (N=21) | Cohort 3: Placebo (N=13) | Cohort 3: Etelcalcetide 5 mg (N=13)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arteriovenous graft site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Placebo (N=4) | Cohort 1: Etelcalcetide 5 mg (N=6) | Cohort 2: Placebo (N=21) | Cohort 2: Etelcalcetide 10 mg (N=21) | Cohort 3: Placebo (N=13) | Cohort 3: Etelcalcetide 5 mg (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.